CLINICAL TRIAL: NCT02861261
Title: Probiotics and BeRberine on the Efficacy and Change of Gut MicrObiota in paTients With Newly Diagnosed Type 2 diabEtes（PREMOTE Study）
Brief Title: A Study on the Efficacy and Gut Microbiota of Berberine and Probiotics in Patients With Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCEMD-20160301
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group A (Experimental)
  Interventions: Drug: 1. Berberine hydrochloride tablets ; 2. ProMetS probiotics powder
- Group B (Experimental)
  Interventions: Drug: 1. Berberine placebo tablets ; 2. ProMetS probiotics powder
- Group C (Experimental)
  Interventions: Drug: 1. Berberine hydrochloride tablets; 2. Probiotics placebo powder
- Group D (Placebo Comparator)
  Interventions: Drug: 1. Berberine placebo tablets; 2. Probiotics placebo powder

INTERVENTIONS:
Drug: 1. Berberine hydrochloride tablets ; 2. ProMetS probiotics powder — 1. 0.6g (6 pills) of Berberine tablets administered twice a day orally before meal ;
  2. 4g (2 strips) of ProMetS probiotics powder administered orally every night
  Arms: Group A
Drug: 1. Berberine placebo tablets ; 2. ProMetS probiotics powder — 1. 6 pills of Berberine placebo tablets administered twice a day orally before meal;
  2. 4g (2 strips) of ProMetS probiotics powder administered orally every night
  Arms: Group B
Drug: 1. Berberine hydrochloride tablets; 2. Probiotics placebo powder — 1. 0.6g (6 pills) of Berberine tablets administered twice a day orally before meal;
  2. 2 strips of probiotics placebo powder administered orally every night
  Arms: Group C
Drug: 1. Berberine placebo tablets; 2. Probiotics placebo powder — 1. 6 pills of Berberine placebo tablets administered twice a day orally before meal;
  2. 2 strips of probiotics placebo powder administered orally every night
  Arms: Group D

SUMMARY:
The purpose of this study is to conduct a multicenter randomized, double-blind, placebo-controlled clinical trial, evaluating the effects and change of gut microbiota after berberine and/or probiotics administration in patients with newly diagnosed type 2 diabetes

DETAILED DESCRIPTION:
In the present study, about 400 newly-diagnosed type 2 diabetes patients will be enrolled from multiple centers in China. Randomisation was computer generated and stratified by age. After screening, eligible subjects will be given Gentamycin Sulfate Sustained-release Tablets 80mg bid po for a week at the washout period, then all participants will be randomly assigned into one of the following four groups: Berberine hydrochloride tablets（0.6g bid po）and ProMetS probiotics powder（4g qN po), Berberine placebo tablets（6 pills bid po) and ProMetS probiotics powder (4g qN po), Berberine hydrochloride tablets（0.6g bid po）and Probiotics placebo powder (2 strips qN po), Berberine placebo tablets（6 pills bid po) and Probiotics placebo powder (2 strips qN po) for 3 months.

The primary objective is to determine whether a combination of probiotics and berberine is preferable to either berberine alone or probiotics alone, in comparison with placebo in improving 1). glycemic control, as measured by change in HbA1c level from baseline to 13-week follow-up, and 2). glycemic control, as measured by change in HbA1c level from baseline to 13-week follow-up in participants aged ≥ 50 years.

Blood, feces and urine samples will be collected before and after treatment. HbA1C, fasting plasma glucose (FPG), postprandial plasma glucose (PPG), GLP-1 , lipids, amino acids, bile acids and other metabolic related components and parameters will be measured. Furthermore, the change of gut microbiota will be evaluated too.

ELIGIBILITY:
Main Inclusion Criteria:

1. Newly diagnosed type 2 diabetes defined as WHO (1999) diagnostic criteria ; Both Genders Eligible;
2. Age: ≥20 and <70 years;
3. BMI: 19.0 ~ 35.0kg/m2;
4. Not receive previously with anti-diabetic agents (oral agents, GLP-1 or insulin);
5. Have at least 2 months of life style intervention to control blood glucose before screening;
6. HbA1c ≥6.5% and ≤10.0%, and fasting plasma glucose≥7.0 mmol/L and ≤13.3mmol/L at screening.

Details please see the study protocol. -

Main Exclusion Criteria:

1. Significant impaired liver function (defined as alanine transaminase (ALT)> 2.5 times upper limit of normal); Impaired renal function (defined as serum-creatinine> 132μmol/L or eGFR <60 mL/min/1.73m2 ); Mental disease, severe infection, severe anemia, neutropenia disease;
2. Other severe heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, defined as New York Heart Association class III or IV;
3. Allergic to gentamicin or other amino glycosides antibiotics;
4. Histories of acute diabetic complications including diabetic ketoacidosis or hyperosmolar hyperglycemic non-ketotic coma within 3 months;
5. Pregnancy;
6. Acute and chronic diarrhea or severe constipation of the digestive tract diseases;
7. Medical history of malignant tumor (except local skin basal cell carcinoma) in the past 5 years;
8. Medical history of intestine, or other digestive tract surgery (such as cholecystectomy) within one year, or other non gastrointestinal surgery within 6 months.

Details please see the study protocol.

-

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 13 weeks

SECONDARY OUTCOMES:
Gut microbiome | 13 weeks
Fasting glucose levels | 13 weeks
2-hour postprandial glucose levels | 13 weeks
Fasting insulin levels | 13 weeks
2-hour postprandial insulin levels | 13 weeks
Serum Triglycerides | 13 weeks
Serum total Cholesterol | 13 weeks
Serum HDL-c | 13 weeks
Serum LDL-c | 13 weeks
Blood metabolomics profile measurement | 13 weeks
  In aid of LC/MS and GC/MS technique, we will measure the metabolomics molecular profile in blood samples before and after treatment. The metabolomics measurement will help to detect the profile of all kinds of bile acid species, lipids species and amino acid species. The composition change of all these biological molecular induced by the treatment is our major interest rather than single molecular quantification
Blood Incretin | 13 weeks
  In aid of multiple ELISA based on xMAP Luminex technology, we will measure gut hormones, including Glp-1, GIP and PYY in ng/ml.
Inflammation markers (hs-CRP, TNF-alfa, IL-6, and IL-8 etc. in ng/ml) | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Y, Gu Y, Ren H, Wang S, Zhong H, Zhao X, Ma J, Gu X, Xue Y, Huang S, Yang J, Chen L, Chen G, Qu S, Liang J, Qin L, Huang Q, Peng Y, Li Q, Wang X, Kong P, Hou G, Gao M, Shi Z, Li X, Qiu Y, Zou Y, Yang H, Wang J, Xu G, Lai S, Li J, Ning G, Wang W. Gut microbiome-related effects of berberine and probiotics on type 2 diabetes (the PREMOTE study). Nat Commun. 2020 Oct 6;11(1):5015. doi: 10.1038/s41467-020-18414-8. PMID 33024120